CLINICAL TRIAL: NCT06948760
Title: Testing a Conversion Factor for a More Rapidly Acting Insulin in an Automated Insulin Delivery System Among Adolescents With T1D [Launchpad Lyumjev]
Brief Title: Testing a Conversion Factor for a More Rapidly Acting Insulin in an Automated Insulin Delivery System Among Adolescents With T1D
Acronym: Lpad Lyumjev
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mark D. DeBoer, MD, MSc., MCR (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Mark D. DeBoer, MD, MSc., MCR, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302376
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Continuous Glucose Monitor (CGM); Tandem t:slim Insulin Pump with Control-IQ Technology (CIQ); Lyumjev insulin; Conversion Factor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lyumjev insulin using settings determined by experimental conversion factor (Experimental): All participants will have a physician-driven insulin Optimization Phase using their home Humalog or Novolog in the Control-IQ control group. After this, participants will have a two-week baseline control phase to assess time-in-range on the optimized insulin settings. Participants will then use Lyumjev insulin for a two-week period with insulin settings determined using the conversion factor.
  Interventions: Device: Control-IQ insulin pump with Lyumjev insulin
- Humalog or Novolog using optimized insulin settings (Active Comparator): All participants will have a physician-driven insulin Optimization Phase using their home Humalog or Novolog in the Control-IQ control group. After this, participants will have a two-week baseline control phase to assess time-in-range on the optimized insulin settings. Participants will then remain on their home Humalog or Novolog for a two-week period using the optimized insulin settings. Each group will have their time-in-range during the randomized phase compared to that during the baseline period.
  Interventions: Device: Control-IQ insulin pump with Humalog or Novolog

INTERVENTIONS:
Device: Control-IQ insulin pump with Lyumjev insulin — Control-IQ insulin pump with insulin using settings determined by experimental conversion factor
  Other Names: Experimental Group
  Arms: Lyumjev insulin using settings determined by experimental conversion factor
Device: Control-IQ insulin pump with Humalog or Novolog — Control-IQ insulin pump with Humalog or Novolog using optimized insulin settings
  Other Names: Control Group
  Arms: Humalog or Novolog using optimized insulin settings

SUMMARY:
A randomized controlled trial of Control-IQ, assessing glycemic control (time-in-range 70-180 mg/dL) for Lyumjev insulin (in which the insulin settings have been determined using an experimental conversion factor) as compared to Humalog or Novolog (using optimized settings)

DETAILED DESCRIPTION:
All participants will have a physician-driven insulin Optimization Phase using their home Humalog or Novolog in the Control-IQ control group. After this, participants will have a two-week baseline control phase to assess time-in-range on the optimized insulin settings. Participants will then be randomized to switch to Lyumjev insulin (with insulin settings determined using the conversion factor) or remain on their home Humalog or Novolog for a two-week period. Each group will have their time-in-range during the randomized phase compared to that during the baseline period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12.0 and ≤22 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. HbA1c >6.5 - 12%
4. Currently using insulin for at least six months
5. Currently using the Tandem t:slim insulin pump with Control-IQ Technology® for at least two months
6. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
7. Access to internet and willingness to upload data during the study as needed, including data generated prior to the start of the study
8. For females, not currently known to be pregnant or breastfeeding
9. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
10. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, prior to the insulin Optimization Phase and for the duration of the study
11. Willingness to use Lyumjev if randomized to the experimental treatment arm
12. Total daily insulin dose (TDD) at least 10 U/day and not more than 100 U/day
13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, sulfonylureas and nutraceuticals)
14. Willingness to eat at least 1 g/kg of carbohydrate per day
15. Willingness to check ketones per study protocol using home urine ketone strips
16. An understanding and willingness to follow the protocol and signed informed consent

Exclusion Criteria:

1. History of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
3. Current HbA1c <6.5 or >12
4. Pregnancy or intent to become pregnant during the trial
5. Currently being treated for a seizure disorder
6. Planned surgery during study duration
7. Need for treatment with oral steroid
8. Treatment with any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and nutraceuticals)
9. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time in Range (70-180 mg/dL) | 14 days
  The primary endpoint of the clinical trial will be the difference in time in range glucose (70-180 mg/dL) by CGM (adjusted for baseline TIR) between those on the Lyumjev conversion factor and those remaining on optimized settings of Humalog/Novolog.

CONTACTS AND LOCATIONS:
Overall Officials: Mark DeBoer, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available after publication of the manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for three years from the publication of the manuscript.
Access Criteria: Data will be available on reasonable request after Data Sharing Agreements have been formulated.
URL: https://med.virginia.edu/diabetes-technology/